CLINICAL TRIAL: NCT06497530
Title: An Exploratory Study of Maintenance Lurbinectedin in Combination With Serplulimab for Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: Maintenance Lurbinectedin in Combination With Serplulimab for Patients With ES-SCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Director, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC-24-02
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): Induction phase：participants will receive Serplulimab on Day 1 of each 21-day cycle in combination with carboplatin on Day 1 and etoposide on Days 1, 2, and 3 of each 21-day cycle for 4 cycles.
  Maintenance phase：participants will receive Serplulimab on Day 1 of each 21-day cycle in combination with Lurbinectedin on Day 1 of each 21-day cycle.
  Interventions: Drug: Serplulimab; Drug: Lurbinectedin; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Serplulimab — Serplulimab will be administered intravenously at a dose of 4.5 mg/kg on Day 1 of each 21-day cycle for 4 cycles in the induction phase.
  Serplulimab will be administered intravenously at a dose of 4.5 mg/kg on Day 1 of each 21-day cycle in the maintenance phase.
Drug: Lurbinectedin — Lurbinectedin will be administered intravenously at a fixed dose of 4 mg on Day 1 of each 21-day cycle in the maintenance phase.
  Other Names: PM01183
Drug: Carboplatin — Carboplatin will be administered according to the standard of care treatment for 4 cycles in the induction phase.
Drug: Etoposide — Etoposide will be administered according to the standard of care treatment for 4 cycles in the induction phase.

SUMMARY:
This is a single-arm, open-lable exploratory study of Lurbinectedin in combination with Serplulimab as maintenance therapy in participants with extensive-stage small-cell lung cancer (ES-SCLC) after first-line induction therapy with carboplatin, etoposide, and Serplulimab. The study consists of 2 phases: an induction phase and a maintenance phase. Participants need to have an ongoing response or stable disease per the Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 criteria after completion of 4 cycles of carboplatin, etoposide, and Serplulimab induction treatment in order to be considered for eligibility screening for the maintenance phase. Eligible participants will receive lurbinectedin plus Serplulimab in the maintenance phase.

ELIGIBILITY:
Inclusion Criteria for the Induction Phase:

* Fully informed about the study and voluntarily signed a written informed consent form, and able to comply with the requirements and restrictions listed in the informed consent form;
* Male or female with age ≥ 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1;
* Histologically or cytologically confirmed diagnosis of extensive-stage small cell lung cancer (ES-SCLC) and has not received any systemic treatment for ES-SCLC;
* At least one measurable lesion (according to RECIST 1.1 criteria);
* Having adequate bone marrow, hepatic, renal and metabolic function, meaning the functional level of the organs meets the following requirements:
* Platelet count (PLT) ≥ 100×10^9/L; Hemoglobin (Hb) ≥ 90 g/L; Absolute neutrophil count (ANC) ≥ 2.0×10^9/L;
* Regardless of whether liver metastasis is present, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0×upper limit of normal (ULN);
* Alkaline phosphatase (ALP) ≤ 5×ULN;
* Total bilirubin (TBIL) ≤ 1.5×ULN, and direct bilirubin ≤ 1.0×ULN;
* Serum creatinine ≤ 1.5×ULN or creatinine clearance rate ≥ 30 mL/min (calculated using the Cockcroft-Gault formula);
* Creatine phosphokinase (CPK) ≤ 2.5×ULN;
* Albumin ≥ 3.0 g/dL.
* Women of childbearing potential(WOCBP) must have a negative serum pregnancy test before enrollment. WOCBP must use effective contraceptive measure during the trial drug treatment and for 6 months after the last administration. Male patients (with partners of WOCBP) must use effective contraceptive measure during the trial drug treatment and for 4 months after the last administration;
* Human immunodeficiency virus (HIV)-negative, with no active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

Exclusion Criteria for the Induction Phase:

* Have a history of central nervous system (CNS) metastasis or related history;
* Have a history of active autoimmune disease or immunodeficiency, or related history;
* Have a history of malignancies other than SCLC within 5 years before enrollment;
* Previous treatment with immune checkpoint inhibitors or lurbinectedin;
* Have a history of idiopathic pulmonary fibrosis or pneumonia, or active pneumonia detected in CT screening;
* Treatment with any other investigational product within 28 days before enrollment.

Inclusion Criteria for the Maintenance Phase:

* Have a continuous response or stable disease according to RECIST 1.1 criteria after 4 cycles of induction therapy;
* Toxicity from the induction therapy phase has recovered to ≤ Grade 1;
* Have sufficient bone marrow and organ function.

Exclusion Criteria for the Maintenance Phase:

* Have a history of central nervous system (CNS) metastasis or related history;
* Has received chest consolidation radiotherapy;
* Severe infection within 2 weeks before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Treatment initiation to the date of first documented disease progression or death whichever occurs first (up to approximately 24 months)
  progression-free survival (PFS) is defined as the time from treatment initiation to the date of first documented disease progression (as assessed according to RECIST v1.1) or death whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Treatment initiation to the date of death from any cause(up to approximately 24 months)
  Overall survival (OS) is defined as the time from treatment initiation to the date of death from any cause.
Objective Response Rate (ORR) | up to approximately 24 months
  Objective response rate (ORR) is defined as the proportion of participants with a complete response（CR） or partial response（PR） according to RECIST v1.1.
Duration of Response (DOR) | up to approximately 24 months
  Duration of Response (DOR) (for participants with a confirmed objective response) is defined as the time from the first occurrence of a documented confirmed objective response until disease progression according to RECIST v1.1 or death from any cause, whichever occurs first.
Percentage of Participants With Adverse Events | up to approximately 24 months
  Percentage of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: chengzhi Zhou, MD, Principal Investigator — Guangzhou Institute of Respiratory Disease

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared